CLINICAL TRIAL: NCT07089212
Title: The Efficacy of Cyclic Compression Cryotherapy Combined With Phased Rehabilitation Training on Lower Limb Functional Recovery in Patients After Total Knee Arthroplasty
Brief Title: Combined Cyclic Compression Cryotherapy and Phased Rehabilitation Training for Recovery After Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KYLL-202502-012-1
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Knee Arthroplasty, Total; Rehabilitation Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rehabilitation treatment. (Active Comparator): The control group underwent a 12-week conventional rehabilitation program, which primarily included muscle strength training, endurance training, proprioception training, and joint range of motion (ROM) exercises. Assessments were conducted at baseline (before treatment), as well as at 2 weeks, 6 weeks, and 12 weeks post-treatment. The evaluated outcomes included knee joint ROM, muscle strength, knee function, pain levels, and activities of daily living (ADL).
  Interventions: Behavioral: Conventional rehabilitation treatment.
- Cyclic cryotherapy combined with staged rehabilitation treatment. (Experimental): The experimental group received cyclic compression cryotherapy combined with phased rehabilitation training in addition to the conventional rehabilitation program, with a total intervention duration of 12 weeks.
  Interventions: Behavioral: Phased Rehabilitation Training; Device: Cyclic Compression Cryotherapy

INTERVENTIONS:
Behavioral: Phased Rehabilitation Training — Rehabilitation is divided into three postoperative phases:
  Early Phase (Weeks 1-2): Focus on edema control, quadriceps activation, and passive/active-assisted range of motion (ROM) exercises.
  Intermediate Phase (Weeks 3-6): Progress to strength training, endurance exercises, and early proprioception drills.
  Late Phase (Weeks 7-12): Advance to functional training , dynamic proprioception, and full ROM restoration.
  Arms: Cyclic cryotherapy combined with staged rehabilitation treatment.
Device: Cyclic Compression Cryotherapy — Initiation: Begin within 24 hours postoperatively. Each session lasts 20-30 minutes, administered 2-3 times daily.
  Procedure: Apply a cryotherapy wrap circumferentially around the knee using a pneumatic compression device, with precise control of pressure and temperature.
  Pressure Settings: Start at Level I-II (low-to-moderate) and adjust incrementally based on patient tolerance.
  Temperature Control: Maintain at 10-12°C.
  Arms: Cyclic cryotherapy combined with staged rehabilitation treatment.
Behavioral: Conventional rehabilitation treatment. — The control group underwent a 12-week conventional rehabilitation program, which primarily included muscle strength training, endurance training, proprioception training, and joint range of motion (ROM) exercises. Assessments were conducted at baseline (before treatment), as well as at 2 weeks, 6 weeks, and 12 weeks post-treatment. The evaluated outcomes included knee joint ROM, muscle strength, knee function, pain levels, and activities of daily living (ADL).
  Arms: conventional rehabilitation treatment.

SUMMARY:
Total knee arthroplasty (TKA) is an effective treatment for severe knee joint diseases; however, postoperative complications such as pain, swelling, and delayed functional recovery remain common challenges. Cyclic compression cryotherapy, which applies alternating cold and pressure to the knee joint, can effectively reduce swelling and alleviate pain. Meanwhile, phased rehabilitation training, tailored to the specific recovery stages post-surgery, facilitates targeted exercise interventions to promote functional restoration of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with knee osteoarthritis (KOA) and within 12 weeks after total knee arthroplasty (TKA).
2. Aged 18-70 years.
3. First-time unilateral TKA (non-revision surgery).
4. Physically and cognitively capable of completing required assessments.
5. Able to fully adhere to the study protocol.
6. Willing to participate in and complete the entire rehabilitation program.
7. No contraindications for surgery or postoperative rehabilitation.
8. Intact cognitive function (able to provide informed consent and follow instructions).
9. Available for all follow-up evaluations.

Exclusion Criteria:

* 1. Severe cardiovascular or cerebrovascular diseases. 2. Neuromuscular impairments affecting the lower limbs. 3. Concurrent hip or ankle joint disorders. 4. Intolerance to pain (unable to tolerate rehabilitation protocols). 5. Primary or metastatic bone tumors. 6. Rheumatoid arthritis (RA) or other systemic inflammatory arthropathies. 7. Severe obesity (BMI ≥35) or malnutrition (clinically diagnosed). 8. Inability to comply with study assessments (e.g., due to cognitive or physical limitations).

  9. Visual dysfunction impairing task performance. 10. Functional impairment of the non-operated limb hindering testing/training. 11. Ankylosing spondylitis (AS). 12. History of allergic hypersensitivity to interventions used in the study. 13. Hemorrhagic predisposition (e.g., coagulation disorders, anticoagulant use).

  14. Active tuberculosis or chronic myelitis. 15. History of substance dependence (e.g., opioids, alcohol). 16. Psychiatric disorders (e.g., schizophrenia, major depression). 17. Severe dysfunction of major organs (e.g., hepatic, renal, pulmonary).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Knee Function Scores | At 6 weeks after completion of treatment.

SECONDARY OUTCOMES:
Range of Motion (ROM) | At 6 weeks after completion of treatment.
Muscle Strength | At 6 weeks after completion of treatment.
Activities of Daily Living (ADLs) | At 6 weeks after completion of treatment.
Visual Analog Scale (VAS) | At 6 weeks after completion of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- 107 Wenhua Xi Road, Ji'nan Shandong 250012, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No